CLINICAL TRIAL: NCT00766506
Title: Comparison of Ionsys and Routine Care With Morphine IV (Intravenous) PCA in the Management of Early Post-operative Mobilisation, Ability to Mobilise and in Time to Fitness For Discharge
Brief Title: An Efficacy and Safety Study to Compare Fentanyl Ionsys and Routine Care With Intravenous (IV) Morphine Patient-controlled Analgesia (PCA) in Participants Who Have Undergone Elective Major Abdominal or Orthopedic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Product class one recall
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015211; FENHYDPAI4012; 2008-000529-20
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-03

CONDITIONS: Pain, Postoperative
Keywords: IONSYS; Fentanyl; Morphine; PCA; Postoperative pain; Mobilization
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl IONSYS (Experimental): Participants will receive 40 microgram (mcg) of fentanyl dose up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 80 doses within a 24 hour period from an Iontophoretic Transdermal System (IONSYS).
  Interventions: Device: Fentanyl IONSYS
- Morphine IV PCA (Active Comparator): Morphine sulphate solution will be administered intravenously (directly into the vein, IV) by a patient-controlled analgesia (PCA) pump using set bolus (a large amount) doses with a fixed lock out period as per physician's discretion (maximum total dose of 20 milligram per 2 hours) for 72 hours.
  Interventions: Device: Morphine IV PCA

INTERVENTIONS:
Device: Fentanyl IONSYS — Participants will receive 40 mcg of fentanyl dose up to a maximum of 240mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 80 doses within a 24 hour period from an Iontophoretic Transdermal System (IONSYS).
  Arms: Fentanyl IONSYS
Device: Morphine IV PCA — Morphine sulphate solution will be administered intravenously (IV) by a patient-controlled analgesia (PCA) pump using set bolus doses with a fixed lock out period as per physician's discretion (maximum total dose of 20 milligram per 2 hours) for 72 hours.
  Arms: Morphine IV PCA

SUMMARY:
The purpose of this study is to evaluate the mobilization characteristics, clinical use, safety and Ease of Care (EOC) of a fentanyl Iontophoretic Transdermal Patient Controlled Analgesia (PCA) system (Ionsys) and morphine intravenous (IV) PCA for management of moderate (medium level of seriousness) to severe (very serious) acute (a quick and severe) pain in participants who have undergone elective major abdominal or orthopedic (pertaining to the bones) surgery.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), multicentre (when more than one hospital or medical school team work on a medical research study), open-label (participants and physicians are told which treatment the participants are receiving), active-controlled (experimental treatment is compared to a standard treatment), parallel group study (a study comparing the response in two or more groups of participants receiving different treatments). The study will consist of 2 phases: screening phase and an open-label treatment phase. The duration of participation in the study for an individual participant will be 72 hours. Eligible participants (who require pain treatment with strong opioids [morphine like medications] for at least 24 hours after an elective spine or elective orthopedic surgery) will be randomly assigned to receive either Ionsys or morphine IV PCA. Participants' safety will be monitored.

ELIGIBILITY:
Inclusion Criteria

* Participants, after an elective major abdominal or orthopedic (pertaining to bones) surgery
* Expected to have acute (a quick and severe form of illness in its early stage) moderate (medium level of seriousness) to severe (very serious) post-operative pain requiring parenteral (administration by injection) opioids (morphine like medication) for at least 24 hours after surgery
* Participants who have undergone General anesthesia (loss of sensation or feeling), spinal anesthesia of less than or equal to 4 hours duration or epidural (outside the spinal cord) anesthesia
* Participants with respiratory rate 10 to 24 breaths per minute
* Participants with a pain score less than or equal to 4 out of 10 on a Numerical Rating Scale (NRS), after titration to comfort with intravenous (IV) morphine Exclusion Criteria
* Surgery secondary to malignancy (cancer or other progressively enlarging and spreading tumor) or trauma (injury)
* History of psychological opioid dependence and/or known or suspected to be opioid dependent
* Severe chronic (lasting a long time) obstructive respiratory symptoms susceptibility to respiratory depression, moderate to severe renal (having to do with the kidney) dysfunction
* Peri-operative administration of opioids other than morphine, fentanyl, sufentanil, alfentanil or remifentanil
* Require high doses of opioids to control their pain (more than 40 milligram morphine IV) during titration to comfort, or more than 6 hours have elapsed since the participant arrived in the recovery room or Monoamine oxidase inhibitors (MAOI) within 14 days pre-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (7):
- United Kingdom (7):
  - Belfast
  - Cardiff
  - Edinburgh
  - Glasgow
  - Liverpool
  - Salford
  - Solihull

REFERENCES:
- See also: Comparison of Ionsys and routine care with morphine IV PCA in the management of early post-operative mobilisation, ability to mobilise and in time to Fitness For Discharge. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=264&filename=CR015211_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl IONSYS: Fentanyl 40 microgram (mcg) per 10 minutes up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 3.2 milligram (80 doses) within 24 hour from an Iontophoretic Transdermal System (IONSYS [a device which uses an electric current to move drug through the skin into the blood]), applied on the intact, non-irritated skin on the chest or upper arm. Duration of study treatment was 72 hours.
- Morphine IV PCA: Morphine sulphate solution administered intravenously (directly into the vein) by a patient-controlled analgesia (PCA) pump using set bolus doses with a fixed lock out period as per physician's discretion (maximum total dose of 20 milligram per 2 hours) for 72 hours.
Period: Overall Study
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Started | 58 | 50
Completed | 53 | 48
Not Completed | 5 | 2
Not completed — Use rescue medication after 3 hours | 3 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl IONSYS: Fentanyl 40 microgram (mcg) per 10 minutes up to a maximum of 240 mcg (6 doses each of 10 minutes duration) per hour but not more than a maximum of 3.2 milligram (80 doses) within 24 hour from an Iontophoretic Transdermal System (IONSYS), applied on the intact, non-irritated skin on the chest or upper arm. Duration of study treatment was 72 hours.
- Total: Total of all reporting groups
Arm/Group | Fentanyl IONSYS | Morphine IV PCA | Total
Number analyzed (Participants) | 58 | 50 | 108
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (12.1) | 58.9 (11.8) | 58.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 25 | 17 | 42

OUTCOME MEASURES:

1. Primary Outcome: Participant's Evaluation of Mean Ability to Mobilize After Surgery
Description: The ability to mobilize was assessed through a combined analysis of participant's responses to the following 3 questions: 1-Because of the system/device, I had to be careful when I used my hands; 2-The system/device made it difficult for me to adjust my position in bed; 3-The system/device interfered with my ability to get out of bed and walk around. All 3 items were scored on a 6-point Likert scale, ranging from "not at all" (score 0) to "a very great deal" (score 5). Total ability to mobilize was assessed as average of 3 scores which range from 0 (best mobility) to 5 (worst mobility).
Time Frame: Hour 72 or early study withdrawal
Population: The intention-to-treat (ITT) population included all participants randomly assigned to study treatment and used the study medication at least once, and who had at least 1 efficacy measure after system application or device enablement (0 hours).
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Units on scale | 0.02 (0.101) [-0.19 to 0.47] | 2.26 (1.146) [1.98 to 2.76]
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Test type: Superiority or Other; p < 0.001, ANCOVA; P-value was calculated from analysis of covariance (ANCOVA), with centre, surgery type and treatment included as covariates in the analysis; Least square mean difference = -2.23, 95% CI 2-sided [-2.55 to -1.91] — Least square mean difference = Least square mean value for Fentanyl IONSYS group minus Least square mean value for Morphine IV PCA group

2. Secondary Outcome: Pain Intensity Numerical Rating Scale (NRS)
Description: Pain intensity NRS measured pain intensity experienced by the participant on a scale, 0 to 10, where 0 means no pain and 10 mean the worst possible pain. Participant's pain intensity was assessed by asking following question to the participant: on a scale 0 to 10 where 0 means no pain, and 10 means the worst possible pain, rate the pain that you have now.
Time Frame: Baseline, Hour 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, study treatment discontinuation or withdrawal, and when participant was fit for discharge (FFD) (assessed up to 91 hours)
Population: The ITT population included all participants randomly assigned to study treatment and used the study medication at least once, and who had at least 1 efficacy measure after system application or device enablement (0 hours). Here 'n' signifies those participants evaluable for this measure at the specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Unit on Scale
  Baseline (n = 58, 49) | 1.2 (1.76) | 1.3 (1.84)
  Hour 1 (n = 58, 48) | 1.6 (2.36) | 1.5 (2.09)
  Hour 2 (n = 57, 49) | 2.2 (2.51) | 2.1 (2.30)
  Hour 3 (n = 57, 48) | 2.7 (2.28) | 2.2 (2.16)
  Hour 4 (n = 57, 47) | 2.9 (2.20) | 2.9 (2.68)
  Hour 5 (n = 58, 46) | 3.1 (2.25) | 2.5 (2.19)
  Hour 6 (n = 55, 46) | 3.1 (2.12) | 2.5 (2.24)
  Hour 8 (n = 54, 44) | 3.0 (1.86) | 2.3 (2.33)
  Hour 12 (n = 48, 40) | 2.5 (2.03) | 1.8 (1.91)
  Hour 24 (n = 52, 34) | 1.5 (1.69) | 1.9 (1.85)
  Hour 48 (n = 13, 6) | 0.6 (0.96) | 1.5 (1.05)
  Hour 72 (n = 3, 2) | 0.7 (1.15) | 0.5 (0.71)
  Study discontinuation or withdrawal (n = 53, 50) | 1.8 (2.66) | 1.6 (1.78)
  FFD (n = 44, 38) | 0.6 (1.06) | 1.3 (1.62)
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; At Hour 24; Test type: Superiority or Other; p = 0.219, ANCOVA; P-value was calculated from ANCOVA, with centre, surgery type and treatment included as covariates in the analysis
Statistical Analysis 2: Comparison: Fentanyl IONSYS vs Morphine IV PCA; At Hour 48; Test type: Superiority or Other; p = 0.299, ANCOVA; P-value was calculated from ANCOVA, with centre, surgery type and treatment included as covariates in the analysis
Statistical Analysis 3: Comparison: Fentanyl IONSYS vs Morphine IV PCA; At study discontinuation or withdrawal; Test type: Superiority or Other; p = 0.136, ANCOVA; P-value was calculated from ANCOVA, with centre, surgery type and treatment included as covariates in the analysis

3. Secondary Outcome: Nurse Ease of Care (EOC) Questionnaire Score
Description: Nurse EOC questionnaire had 22 items and covered 3 aspects of care delivery associated with acute care pain management systems: time, bothersome and satisfaction. Items were scored on a 6-point Likert scale, ranging from 'not at all' (Score 0) to 'a very great deal' (score 5). The total score was calculated as the mean of the non-missing items for all the questions.
Time Frame: When participant was fit for discharge (FFD) (assessed up to 91 hours)
Population: The ITT population included all participants randomly assigned to study treatment and used the study medication at least once, and who had at least 1 efficacy measure after system application or device enablement (0 hours).
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on scale
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Units on scale | 0.28 (0.399) [0.07 to 0.49] | 0.80 (0.547) [0.55 to 1.05]
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Test type: Superiority or Other; p < 0.001, ANCOVA; P-value was calculated from ANCOVA, with centre, surgery type and treatment included as covariates in the analysis; Least square mean difference = -0.52, 95% CI 2-sided [-0.74 to -0.30] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Patient Global Assessment (PGA) of Method of Pain Control
Description: The assessment consist of a categorical evaluation (poor, fair, good or excellent) of the method of pain control by asking following question from the participant: "Overall, would you rate this PCA (participant controlled analgesia) method of pain control as being poor, fair, good, or excellent?"
Time Frame: Hour 72 or early study withdrawal
Population: The ITT population included all participants randomly assigned to study treatment and used the study medication at least once, and who had at least 1 efficacy measure after system application or device enablement (0 hours). Here 'N' (number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Number; unit: Participants
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 49
Participants
  Poor | 5 | 1
  Fair | 1 | 6
  Good | 21 | 23
  Excellent | 31 | 19
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Test type: Superiority or Other; p = 0.131, Mantel Haenszel; P-value was calculated from a Mantel-Haenszel Chi-Squared test; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.84 to 3.92]

5. Secondary Outcome: Time to Fit For Discharge (FFD)
Description: Participants were assessed for fulfilling the following FFD criteria: 1- Retaining fluids and food; 2- Passing urine without the aid of a catheter; 3- Bowel sounds and/or opening; 4- Cardiovascular stability; 5- Respiratory stability; 6- No post-operative wound complications; 7- Pain adequately controlled with oral analgesia only; 8- Adequately mobile according to locally acceptable standards for mobility for surgery type and pre-operative expectations. The FFD criteria were answered on a "Yes" or "No" basis. When all criteria were answered as Yes, participant was considered to be FFD.
Time Frame: When participant was FFD (assessed up to 91 hours)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Hours | 70.08 [65.50 to 72.25] | 71.21 [67.42 to 90.77]
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Test type: Superiority or Other; p = 0.342, Log Rank; P-value was calculated from a log-rank test stratified for surgery type

6. Other Pre Specified Outcome: Time to Actual Discharge
Description: The time from baseline to the time at which the participant was actually discharged from ward care was recorded as time to actual discharge.
Time Frame: When participant was actually discharged from ward care (assessed up to 258.5 hours)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Hours | 91.44 [75.33 to 96.50] | 94.61 [76.77 to 96.08]
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Test type: Superiority or Other; p = 0.836, Log Rank; P-value was calculated from a log-rank test stratified for surgery type

7. Secondary Outcome: Number of Participants Who Require Rescue Medication
Description: Rescue medication was defined as a fast-acting medication given besides the study drug that could alleviate pain quickly, but the effects were not long lasting. Morphine was given intravenously as rescue medication for all participants randomly assigned to either treatment group.
Time Frame: Baseline up to Hour 3
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Participants | 10 | 2
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Test type: Superiority or Other; p = 0.029, Chi-squared; Odds Ratio (OR) = 5.00, 95% CI 2-sided [1.04 to 24.03]

8. Secondary Outcome: Number of Participants Who Require Concomitant Antiemetic Medication
Description: Antiemetic medicines are the drugs which prevent vomiting.
Time Frame: Baseline up to end of study treatment (Hour 72)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Participants
  Dexamethasone | 1 | 0
  Cyclizine | 19 | 20
  Metoclopramide | 0 | 3
  Domperidone | 1 | 0
  Ondansetron | 11 | 12
  Granisetron | 2 | 2
  Mentha X Piperita | 0 | 1

9. Secondary Outcome: Number of Participants Who Require Concomitant Non-opioid Analgesics
Description: Non-opioid analgesics are non morphine like medications used to get relieve from pain.
Time Frame: Baseline up to end of study treatment (Hour 72)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Participants
  Paracetamol | 39 | 28
  NSAID's | 31 | 20
Statistical Analysis 1: Comparison: Fentanyl IONSYS vs Morphine IV PCA; Paracetamol: P-value was calculated using Chi-squared test; Test type: Superiority or Other; p = 0.230, Chi-squared; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.74 to 3.53]
Statistical Analysis 2: Comparison: Fentanyl IONSYS vs Morphine IV PCA; NSAID's: P-value was calculated using Chi-squared test; Test type: Superiority or Other; p = 0.163, Chi-squared; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.80 to 3.70]

10. Other Pre Specified Outcome: Number of Participants Facing Technical Failure of the Device
Description: Technical failure was defined as malfunctioning or failure of device to work appropriately.
Time Frame: Baseline up to end of study treatment (Hour 72)
Population: Safety population included all participants randomly assigned to study treatment and who used either of the study treatment at least once.
Measure: Number; unit: Participants
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Number analyzed (Participants) | 58 | 50
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From the time a signed informed consent form was obtained until the participant was discharged from ward care
Arm/Group | Fentanyl IONSYS | Morphine IV PCA
Serious Adverse Events (participants affected / at risk) | 1/58 | 2/50
Other Adverse Events (participants affected / at risk) | 40/58 | 38/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl IONSYS (N=58) | Morphine IV PCA (N=50)
Wound infection (Infections and infestations) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl IONSYS (N=58) | Morphine IV PCA (N=50)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Bradycardia (Cardiac disorders) | 4 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 19 | 13
Vomiting (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Application site erythema (General disorders) | 5 | 0
Pain (General disorders) | 5 | 0
Application site vesicles (General disorders) | 2 | 0
Catheter Site pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Inflammation of wound (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1
Bladder injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 4 | 4
Electrocardiogram abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 6
Syncope vasovagal (Nervous system disorders) | 3 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 4
Haematuria (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Perioperative analgesia (Surgical and medical procedures) | 1 | 0
Spinal anaesthesia (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 14 | 13
Hypertension (Vascular disorders) | 3 | 1
Haematoma (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Wound haemorrhage (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was temporarily stopped due to an issue with a batch of drug outside the study and later permanently stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less